CLINICAL TRIAL: NCT03372187
Title: Pilot and Feasibility Trial of a Telehealth Dietary Intervention for MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: pending
Record Dates: First submitted 2017-11-17; First posted 2017-12-13 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: diet; MS; Telehealth
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: All 20 participants will be placed into the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DIET-MS (Experimental): This group will follow a low glycemic load diet plan prescribed to them by a health coach and will receive information on exercise as well. This group will have weekly calls with the telehealth coach and will be provided access to the eHealth platform.
  Interventions: Behavioral: DIET-MS

INTERVENTIONS:
Behavioral: DIET-MS — Following the completion of testing, all 20 participants will be placed into the DIET-MS group and will follow the prescribed diet plan for 12 weeks. At the end of the 12 weeks, the participants will return to complete follow up testing.

SUMMARY:
This project aims to determine the feasibility of delivering a comprehensive behavioral lifestyle intervention including dietary and exercise components via an evidence based, internet-delivered telehealth coaching platform. Further, investigators will gather preliminary data on the change in multiple sclerosis clinical outcomes and cardiometabolic risk factors after participation in the intervention. The outcomes will inform the design of a larger randomized controlled trial.

ELIGIBILITY:
Inclusion criteria:

1. Relapsing-Remitting Multiple Sclerosis
2. On disease modifying treatment for 6 months
3. No relapse within the previous 30 days
4. Self-identify as not currently meeting recommendations for healthy diet and physical activity
5. Ambulatory with or without assistance
6. Reliable access to the internet via computer or smartphone
7. Be responsible for their personal food preparation or have input into the food prepared for them

Exclusion criteria

1. Unstable cardiovascular disease
2. Unstable renal disease
3. Unstable pulmonary disease
4. Physician does not approve participation

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dietary adherence | 1 year
  Assessed by number of dietary behavior changes made
Physical activity adherence | 1 year
  Assessed by number of physical activity behavior changes made

SECONDARY OUTCOMES:
Feasibility of intervention implementation | 1 year
  Assessed by number of sessions attended

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No